CLINICAL TRIAL: NCT06658418
Title: Erector Spinae Plane Block with Dexmedetomidine and Bupivacain Versus Dexamethasone and Bupivacain for Postoperative Analgesia in Patients Undergoing Abdominal Surgeries
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Loay Gamal (Other)
Responsible Party: Sponsor-Investigator, Loay Gamal, LGamal, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: erector spinae plane block
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Analgesia, Postoperative
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dexmedetomidine combined with bupivacaine (Active Comparator): use for Dexmedetomidine and bupivacain for erector spinae plane block
  Interventions: Procedure: Erector Spinae Plane Block
- dexamethasone combined with bupivacaine (Experimental): use of dexamethasone combined with bupivacaine for erector spinae plane block
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — dexmedetomidine combined with bupivacaine versus dexamethasone combined with bupivacaine for ultrasound-guided ESPB for postoperative pain control in patients scheduled for abdominal surgeries.

SUMMARY:
To compare the analgesic effect of dexmedetomidine combined with bupivacaine versus dexamethasone combined with bupivacaine for ultrasound-guided ESPB for postoperative pain control in patients scheduled for abdominal surgeries

ELIGIBILITY:
Inclusion Criteria:

Age :18 years old and older. Patients undergoing open abdominal surgery.

Exclusion Criteria:

1. Patient refusal
2. known sensitivity or contraindication to any of study drugs
3. contraindications for local anesthesia
4. Patients with local infection at site of puncture
5. uncooperative patients
6. history of psychological disorders or chronic pain and significant liver or renal disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
VAS score | at 30 minutes, 2, 4, 6, 8, 12, 16, 20, and 24 hours postoperative.
  pain intensity using VAS score

SECONDARY OUTCOMES:
the time for requirement of first morphine dose | at 30 minutes, 2, 4, 6, 8, 12, 16, 20, and 24 hours postoperative.
  the time for requirement of first morphine dose (hours)

REFERENCES:
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538